CLINICAL TRIAL: NCT05798468
Title: Comparative Study of Augmented Reality in the Teaching of Health University Students.
Brief Title: Effectiveness of Augmented Reality in the Teaching of Health University Students.
Acronym: AR2022
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Collaborators: Alejandro Vega Morales (Unknown); María Jesús Viñolo Gil (Unknown)
Responsible Party: Principal Investigator, Rocío Martín Valero, PhD, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: UMA_Aumentaty 2022
Record Dates: First submitted 2022-11-25; First posted 2023-04-04 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Education
Keywords: Augmented reality; Usability; Competencies
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Both the teacher who will perform the intervention and the evaluator of the study will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): There will be two control groups. One control group will belong to the University of Malaga and the other will belong to the University of Cadiz. This group will follow the traditional teaching method. The total sample of the group will be approximately 96 students, ensuring a homogeneous distribution between the two groups.
  Interventions: Other: Control group
- Experimental group (Experimental): There will be two experimental groups. One experimental group will belong to the University of Malaga and will use augmented reality using Zapworks software while the other experimental group will belong to the University and will use the Aumentaty platform. The sample will be made up of approximately 107 students, ensuring a homogeneous distribution between the two groups. Both the software and the platform mentioned above will work with augmented reality in the educational field, in this case in the university environment.
  Interventions: Other: Augmented reality

INTERVENTIONS:
Other: Augmented reality — The intervention will be carried out in the Physiotherapy Degree of the Universities of Malaga and Cadiz. It will consist of the use of software and a platform that works with augmented reality. Previously a study of the demographic variable of the population that conforms the study will be carried out. During the intervention, teaching will be carried out with the support and enhancement of the use of augmented reality through Zapworks and Aumentaty. A study and analysis of the variables of the qualifications and usability of the study population will be carried out. For the qualification variable, the academic performance of the students will be taken into account and for the usability variable, the System Usability Scale will be used. Subsequently, an analysis and interpretation will be carried out to assess the correlation between both variables.
  Arms: Experimental group
Other: Control group — Traditional education will be carried out
  Arms: Control group

SUMMARY:
The exponential growth of new technologies has meant that the educational field has had to update itself. From the educational point of view, there are some studies that have promoted the implementation of new technologies. These facts have raised the need to implement augmented reality in the university environment, especially among students of health sciences. The use of augmented reality can mean a new approach to teaching by teachers and better learning by students. Objetive: To compare the degree of usability of the two augmented reality applications and to analyse the academic performance of the control group and the experimental group at the Universities of Cadiz and Malaga. The existence of significant differences and relationships between the two variables will be observed.

DETAILED DESCRIPTION:
This research has followed the SPIRIT statement and the ethical and legal aspects of the Principles of the Declaration of Helsinki. An intervention was carried out using two augmented reality applications in the subject of General Procedures in Physiotherapy II at the Universities of Malaga and Cadiz.

ELIGIBILITY:
Inclusion Criteria:

* Students who belong to the degree of Physiotherapy and who are enrolled in the subject General Procedures in Physical Therapy II.

Exclusion Criteria:

* Non-university students.
* Non-university students from outside the health care field.

Ages: 17 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 203 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Demographic variables | 3 months
  This variable allows us to know the age and gender of the study population. This will allow us to know the homogeneity and the average of the groups that will make up the study. The data of this variable will be obtained through the interview process in the selection and agreement to belong to the study.
Rating variable | 3 months
  This variable will allow us to know the academic performance of the population. An analysis and interpretation of the results of this variable will be carried out individually, that is to say, the results pertaining to the population of the University of Malaga and Cadiz will be observed.
  The unit of measurement will be the academic performance of the students, which will be determined by the teaching tests that evaluate the comprehension, understanding and learning of the knowledge imparted in the subject. The higher the scores or the better the results in the teaching tests, the higher the academic performance, and on the contrary, the lower the scores or the worse the results in the teaching tests, the lower the academic performance.
Usability variable | 3 months
  This variable will take into account the use of Zapworks software and the Aumentaty platform in the study population. The System Usability Scale will be used for data collection. The analysis and interpretation of the data will be carried out individually, i.e., it will be carried out at the universities of Malaga and Cadiz.
  The following questions are the original ones, taken from the original test on The scale consists of 10 questions and each of them can be scored from 1 to 5, where 1 means total disagreement and 5 means total agreement. To obtain the measurement we will add the results obtained by the scale. For this, the odd questions (1,3,5,7 and 9) will take the value assigned by the user and one point will be subtracted. The even numbered questions will be five minus the assigned value. Once the final number is obtained, it will be multiplied by 2.5. The higher the score, the higher the usability and conversely, a lower score will indicate a lower usability.

SECONDARY OUTCOMES:
Correlatión between usability and rating variable | 3 months
  This variable will allow us to perform an interpretation and analysis that will allow us to know whether or not there is a correlation between the rating variable (which measures the students' academic performance) and usability (data that will be obtained from the usability scale). The measurement of the correlation between both variables will be done with Spearman's correlation coefficient, which will determine the existence of a correlation between the two main variables.

CONTACTS AND LOCATIONS:
Overall Officials: Rocío Martín Valero, PhD, Principal Investigator — University Malaga
Locations (1):
- Rocío Martín-Valero, Málaga, Spain

REFERENCES:
- See also: This link takes you directly to the Zapworks software home page. — https://zap.works/